CLINICAL TRIAL: NCT00213486
Title: Weekly Cisplatin/Irinotecan and Radiotherapy in Patients With Locally Advanced Esophageal Cancer: Phase II Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001/141/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2005-09

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Irinotecan

INTERVENTIONS:
Drug: irinotecan

SUMMARY:
The standard non surgical therapy of locally advanced esophageal cancer is based on a definitive concurrent chemoradiotherapy regimen with fluorouracil and cisplatin. One of the alternative regimen which is being studied is the combination of a weekly cisplatin and irinotecan schedule with radiotherapy. This multicentric phase II clinical trial primarily aimed to evaluate the clinical complete response rate and secondary objectives were toxicity profile and survival.

DETAILED DESCRIPTION:
Chemotherapy with weekly cisplatin 30 mg/m2 AND Irinotecan 60 mg/m2 was administered at days1,8,22,29 and concurrently with radiotherapy t days 43,50,64,71. Radiotherapy was delivered day 43 to 75 with 50Gy in 25 fractions/5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* esophageal carcinoma (squamous cell or adenocarcinoma) histologically confirmed
* performance status <OR=2 (ECOG)
* caloric intake>1500 KCal/d
* serum albumin >32 gr/l
* serum creatinine<120 microgr/l
* total serum bilirubin < 1.5 mg/ml
* no prior chemotherapy or radiotherapy or surgery for esophageal neoplasm
* no prior history of malignancy other than cell carcinoma of the skin, in siyu cervical carcinoma, or head and neck carcinoma with complete response since 3 years
* written informed consent

Exclusion Criteria:

* Gilbert's syndrome
* cardiac disease as NYHA class 3 or 4
* myocardial infarction within the previous 6 months
* metastatic disease
* histologically proved invasion of tracheobronchial tree
* metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43
Dates: Start 2002-06; Study Completion 2004-12

PRIMARY OUTCOMES:
clinical complete response defined as no tumor detectable on esophagus endoscopy and no appearance of distant metastasis on CT scan

SECONDARY OUTCOMES:
toxicity profile
overall survival rate at one and two years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MICHEL, MD, Principal Investigator — Federation Francophone de Cancerologie Digestive
Locations (1):
- CHU de Rouen, Rouen, France